CLINICAL TRIAL: NCT00756132
Title: Role of Inflammatory Markers in Predicting Disease Recurrency and Cognitive Performance in Women With High Risk and Locally Advanced Breast Cancer
Brief Title: Using Bio Markers to Predict Disease Recurrence and Cognitive Function in High Risk Breast Ca
Acronym: Cyto-Cog
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: BernLCyto-Cog
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Locally Advanced Breast Cancer; Breast Cancer
Keywords: Breast; Neoplasm; Locally Advanced; Stage IV; Stage III; Cognitive Function; Cytokines; Inflammatory; Node positive
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Bloods Only (B): Women aged 18-65 years with a newly diagnosed locally advanced or high risk operable breast cancer
- A-Cog: Women aged 18-65 years newly diagnosed with LABC/high risk who are willing and able to complete cognitive testing.
- Control (C): Healthy women aged 18-65 years who are willing and able to complete cognitive testing.
- A1-Cog: Women newly diagnosed locally advanced or high risk breast cancer that qualify for cognitive testing but have a condition related to elevated serum levels of cytokines or other inflammatory markers.

SUMMARY:
Women with breast cancer undergo treatments that decrease the chance of recurrence of cancer, but are associated with several side effects, including declines in memory and attention and other thinking abilities. The causes of these declines are not known. However, we know that (i) people with cancer may have high levels of molecules in the blood (cytokines) that reflect inflammation; (ii) injection of cytokines into animals, and their use to treat some human diseases, can lead to decreased memory and attention; and (iii) in some advanced cancers cytokines predict disease outcome. This longitudinal study evaluates the relation of cytokines to decreased thinking abilities and to disease outcome over time. Results of this study may help develop interventions to prevent or minimize cognitive decline and identify women who are at high risk for recurrence, and such information could be used in treatment decisions and in the development of new treatment options.

DETAILED DESCRIPTION:
SCIENTIFIC ABSTRACT Background: Women with locally advanced breast cancer (LABC), and women with high risk (T2-3/N+4, triple negative) yet operable breast cancer, undergo combined treatment including chemotherapy, surgery, irradiation, and hormonal treatment. These treatments decrease the chance of recurrence of cancer, but are associated with several side effects, including cognitive difficulties. About one third of breast cancer patients treated with chemotherapy report sustained decline in thinking abilities ('chemofog') after treatment. The causes for cognitive declines are not known. However there is recent information that: (i) people with cancer may have high levels of cytokines and other inflammatory molecules in the blood; (ii) injection of cytokines into animals, and their use to treat some human diseases, can lead to problems in memory and other cognitive abilities; (iii) some survivors of breast cancer have very high cytokine levels with no evidence that their cancer is still active and (iv) in some advanced cancers different cytokines and other inflammatory markers have prognostic information for disease outcome. Genetic polymorphisms of neuronal proteins (APOe, BDNF, COMT) are predictive for cognitive decline in non-cancer population). Objective: This longitudinal study will determine whether serum levels of cytokines and other inflammatory markers are related to 1) cognitive dysfunction; and 2) recurrence of disease in women with LABC/High Risk. Method: In 120 women with LABC/High risk relation of cytokines and inflammatory markers to cancer recurrence will be evaluated; blood will be drawn pre-chemotherapy, pre-surgery and then 1 and 2 years after diagnosis. In a subset of 60 women with LABC/high risk, cognitive performance will be evaluated at similar times as blood will be drawn. Similarly, a control group of 60 healthy women will be evaluated for cytokines and cognitive performance. We will also evaluate the predictive role of polymorphisms in genes encoding the neuronal proteins APOe, BDNF, and COMT for cognitive impairment. Data Analysis: The impact of cytokine levels and other inflammatory markers on cognitive performance over time will be evaluated using mixed model regression. Multivariate model will be applied to assess the impact of LABC/high risk and chemotherapy on cognitive functions. Cox proportional-hazard model will evaluate the relationship of cytokines and other blood markers on Time-To-Progression to identify variables that predict reoccurrence. Hypotheses: Cytokines and inflammatory markers are related to cognitive impairment and in disease outcome in women with locally advanced and high risk operable breast cancers. Genetic polymorphisms of neuronal proteins (APOe, BDNF, and COMT) are predictive for increased cognitive decline after diagnoses and treatment of these cancers. Implications: Increased knowledge about the causes of cognitive problems in women with breast cancer should allow development of strategies to prevent or minimize these unpleasant symptoms. Cytokines and other biomarkers might be predictive for disease outcome in women with breast cancer and used in tailoring of adjuvant treatment and as potential targets in development of new therapies.

ELIGIBILITY:
Inclusion Criteria:

* (i) women age 18-65, (ii) for group A: women with histologically confirmed invasive breast cancer that is locally advanced (inflammatory and non-inflammatory LABC - any T3-T4 M0 and/or N2-3 M0 stages)
* women 18-65 with histologically confirmed high risk operable breast cancer (T2 and/or N+ M0 endocrine unresponsive breast cancers (ER- and PR-). and HER-2-/+, or any operable breast cancer with ≥ 4 involved axillary lymph nodes
* for group B (healthy controls): healthy women 18-65

Exclusion Criteria:

* (i) conditions that are associated with elevated serum levels of cytokines and other inflammatory markers (major inflammatory, chronic infectious or autoimmune systemic disease, cardiovascular disease, diabetes mellitus type I and II), or (ii) any concomitant or prior malignant disease. Those recruited for evaluation on cognitive functions will also be excluded for (iii) major pre-existing psychiatric history (including depression), dementia, alcohol abuse, or currently using a psychotropic medication that might lead to cognitive problems, (iv) insufficient English skills to comprehend the task instructions, and (v) impaired colour vision for reasons related to some of the test stimuli and tasks.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women ages 18-65 with a newly diagnosed locally advanced breast cancer and healthy women ages 18-65.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2012-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Cognitive performance expressed by raw scores, T and Z scores | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lori Bernstein, PhD, Principal Investigator — University Health Network, Princess Margaret Hospital; Bostjan Seruga, MD, Principal Investigator — PMH UHN
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada